CLINICAL TRIAL: NCT02722668
Title: Transplantation of Umbilical Cord Blood From Unrelated Donors in Patients With Hematological Diseases Using a Non-Myeloablative Preparative Regimen
Brief Title: UCB Transplant for Hematological Diseases Using a Non Myeloablative Prep
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015LS149; MT2015-17 (Other: University of Minnesota Clinical Trials Office)
Record Dates: First submitted 2016-03-24; First posted 2016-03-30 (Estimated); Results first posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Acute Leukemia; Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia/Lymphoma; Burkitt's Lymphoma; Natural Killer Cell Malignancies; Chronic Myelogenous Leukemia; Myelodysplastic Syndrome; Large-cell Lymphoma; Hodgkin Lymphoma; Multiple Myeloma; Relapsed Chronic Lymphocytic Leukemia; Relapsed Small Lymphocytic Lymphoma; Marginal Zone B-cell Lymphoma; Follicular Lymphoma; Lymphoplasmacytic Lymphoma; Mantle-cell Lymphoma; Prolymphocytic Leukemia; Bone Marrow Failure Syndromes; Myeloproliferative Neoplasms/Myelofibrosis; Biphenotypic/Undifferentiated/Prolymphocytic Leukemias; MRD Positive Leukemia; Leukemia or MDS in Aplasia; Relapsed T-Cell Lymphoma; Relapsed Multiple Myeloma; Plasma Cell Leukemia
Keywords: AML; ALL; CML; CLL; SLL
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Myelodysplastic Syndromes; Dendritic Cell Sarcoma, Interdigitating; Hodgkin Disease; Multiple Myeloma; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Prolymphocytic; Bone Marrow Failure Disorders; Myeloproliferative Disorders; Primary Myelofibrosis; Leukemia; Lymphoma, T-Cell; Leukemia, Plasma Cell | interventions — fludarabine; fludarabine phosphate; Cyclophosphamide; Mycophenolic Acid; Sirolimus; Whole-Body Irradiation; Antilymphocyte Serum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- No Anti-thymocyte Globulin (ATG) (Experimental): Hematologic malignancy patients who have received a previous autologous transplant or ≥ 2 cycles of multi-agent chemotherapy within the 3 months previous to umbilical cord blood transplantation.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Drug: MMF; Drug: Sirolimus; Radiation: TBI; Biological: Umbilical cord blood cell infusion
- Anti-thymocyte Globulin (ATG) (Experimental): Hematologic malignancy patients who have not been treated with prior autologous transplant or ≤ 1 cycle of chemotherapy in the 3 months previous to umbilical cord blood transplantation, should receive Anti-thymocyte Globulin (ATG) as part of their conditioning regimen.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Drug: MMF; Drug: Sirolimus; Radiation: TBI; Biological: Umbilical cord blood cell infusion; Biological: ATG

INTERVENTIONS:
Drug: Fludarabine — Both Arms: 30 mg/m^2 IV over 1 hour Day -6 to Day -2
  Other Names: Fludara
Drug: Cyclophosphamide — Arm 1: 50 mg/kg IV over 2 hours Day -6
  Other Names: Cytoxan
Drug: MMF — Both Arms:
  Mycophenolate mofetil (MMF) 3 gram/day IV/PO for patients who are ≥ 40 kg divided in 2 or 3 doses. In obese patients (>125% IBW) 15 mg/kg every 12 hours may be considered. Pediatric patient (<40 kilograms) will receive MMF at the dose of 15 mg/kg/dose every 8 hours beginning Day -3. MMF dosing will be monitored and altered as clinically appropriate based on institutional guidelines. Patients will be eligible for MMF dosing and pharmacokinetics studies.
  Stop MMF at Day +30 or 7 days after engraftment, whichever day is later, if no acute graft versus host disease (GVHD). (Definition of engraftment is 1st day of 3 consecutive days of absolute neutrophil count [ANC) ≥ 0.5 x 109 /L]). If no donor engraftment, do not stop MMF.
  Other Names: Mycophenolate Mofetil
Drug: Sirolimus — Both Arms:
  Adult Dosing: Sirolimus will be administered starting at Day -3 with 8-12 mg oral loading dose followed by single dose 4 mg/day with a target serum concentration of 3 to 12 mg/mL by high-performance liquid chromatography (HPLC) and will be monitored per institutional guidelines. In the absence of acute GVHD sirolimus may be tapered starting at Day +100 and eliminated by Day +180 post-transplantation.
  Pediatric Dosing: Sirolimus will be administered starting on Day -3 with an oral loading dose of 10 mg followed by maintenance dosing of 2.5 mg/m^2/day (Maximum total daily dose of 4mg) as per institutional guidelines. Target serum concentration goals are 3 to 12 mg/mL by high-performance liquid chromatography (HPLC) and will be monitored per institutional guidelines.
  Other Names: Rapamycin
Radiation: TBI — Both Arms: 200 cGy on Day -1
  Other Names: Total body irradiation
Biological: Umbilical cord blood cell infusion — Both Arms: Day 0
  Other Names: UCB
Biological: ATG — Arm 2: 15 mg/kg IV every 12 hours Day -6 to Day -4
  Other Names: Anti-thymocyte Globulin
  Arms: Anti-thymocyte Globulin (ATG)

SUMMARY:
This is a phase II trial using a non-myeloablative cyclophosphamide/ fludarabine/total body irradiation (TBI) preparative regimen with modifications based on factors including diagnosis, disease status, and prior treatment. Single or double unit selected according to current University of Minnesota umbilical cord blood graft selection algorithm.

ELIGIBILITY:
Inclusion Criteria:

* Age, Performance Status, and Graft Criteria

  * <70 years of age with no matched 5/6 or 6/6 sibling donor - patients ≥ 70 and ≤ 75 years of age may be eligible if they have a Co-Morbidity score ≤ 2 (http://www.qxmd.com/calculate-online/hematology/hct-ci)
  * Karnofsky score ≥ 70% (≥ 16 years) or Lansky score ≥ 50 (< 16 years)
  * UCB graft selected according to current University of Minnesota umbilical cord blood graft selection algorithm
* Eligible Diseases All diseases listed below are advanced hematologic malignancies not curable by conventional chemotherapy. Responses to conventional treatment range from zero to 30% but are typically short lived.

  * Acute Leukemias: Must be in remission by morphology (<5% blasts). Note cytogenetic relapse or persistent disease without morphologic relapse is acceptable. Also a small percentage of blasts that is equivocal between marrow regeneration vs. early relapse are acceptable provided there are no associated cytogenetic markers consistent with relapse.

    * Acute Myeloid Leukemia (AML) and related precursor neoplasms: 2nd or greater complete remission (CR); first complete remission (CR1) in patients > 60 years old; CR1 in ≤ 60 years old that is NOT considered as favorable-risk. Favorable risk AML is defined as having one of the following:

      * t(8,21) without cKIT mutation
      * inv(16) or t(16;16) without cKIT mutation
      * Normal karyotype with mutated NPM1 and wild type FLT-ITD
      * Normal karyotype with double mutated CEBPA
      * Acute prolymphocytic leukemia (APL) in first molecular remission at the end of consolidation
    * Acute lymphoblastic leukemia (ALL)/lymphoma: second or greater CR; CR1 unable to tolerate consolidation chemotherapy due to chemotherapy-related toxicities; CR1 high-risk ALL. High risk ALL is defined as having one of the following:

      * Evidence of high risk cytogenetics, e.g. t(9;22), t(1;19), t(4;11), other MLL rearrangements, IKZF1
      * 30 years of age or older at diagnosis
      * White blood cell counts of greater than 30,000/mcL (B-ALL) or greater than 100,000/mcL (T-ALL) at diagnosis
      * CNS leukemia involvement during the course of disease
      * Slow cytologic response (>10% lymphoblasts in bone marrow on Day 14 of induction therapy)
      * Evidence of persistent immonophenotypic or molecular minimal residual disease (MRD) at the end of induction and consolidation therapy
  * Biphenotypic/Undifferentiated/Prolymphocytic Leukemias in first or subsequent CR
  * Chronic myelogenous leukemia in chronic or accelerated phase, or CML blast crisis in morphological remission (<5% blasts): Chronic phase patients must have failed at least two tyrosine kinase inhibitors, been intolerant to all available TKIs, or have T315I mutation.
  * Myelodysplastic syndrome: IPSS INT-2 or High Risk; R-IPSS High or Very High; WHO classification: RAEB-1, RAEB-2; Severe Cytopenias: ANC < 0.8, Anemia or thrombocytopenia requiring transfusion; Poor or very poor risk cytogenetics based on IPSS or R-IPSS definitions; therapy-related MDS. Blasts must be < 5% by bone marrow aspirate morphology. If ≥5% blasts, patient requires chemotherapy for cytoreduction to <5% blasts prior to transplantation.
  * MRD positive leukemia (AML, ALL or accelerated/blast phase CML). Selected patients in morphologic CR, but with positive immunophenotypic (flow cytometry) or molecular evidence of MRD may be eligible if recent chemotherapy has not resulted in MRD negative status.
  * Leukemia or MDS in aplasia. These patients may be taken to transplant if after induction therapy they remain with aplastic bone marrow and no morphological or flow-cytometry evidence of disease ≥ 28 days post-therapy. These high risk patients will be analyzed separately.
  * Burkitt's lymphoma in CR2 or subsequent CR
  * Relapsed T-Cell Lymphoma that is chemotherapy sensitive in CR/PR that has failed or ineligible for an autologous transplant.
  * Natural killer cell malignancies
  * Large-cell lymphoma, Hodgkin lymphoma and multiple myeloma with chemotherapy sensitive disease who are ineligible for an autologous transplant.
  * Relapsed Chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL), marginal zone B-cell lymphoma, follicular lymphoma which have progressed within 12 months of achieving a partial or complete remission. Patients who had remissions lasting > 12 months, are eligible after at least two prior therapies. Patients with bulky disease should be considered for debulking chemotherapy before transplant. Patients with refractory disease are eligible, unless bulky disease and an estimated tumor doubling time of less than one month.
  * Lymphoplasmacytic lymphoma, mantle-cell lymphoma, prolymphocytic leukemia are eligible after initial therapy if chemotherapy sensitive.
  * Relapsed Multiple Myeloma that is chemotherapy sensitive and has failed or ineligible for an autologous transplant.
  * Plasma Cell Leukemia after initial therapy if achieved at least in partial remission; or relapsed and achieved subsequent remission (CR/PR)
  * Acquired Bone marrow failure syndromes, except for Fanconi anemia
  * Myeloproliferative Neoplasms/Myelofibrosis
  * Other Leukemia Subtypes: A major effort in the field of hematology is to identify patients who are of high risk for treatment failure so that patients can be appropriately stratified to either more (or less) intensive therapy. This effort is continually ongoing and retrospective studies identify new disease features or characteristics that are associated with treatment outcomes. Therefore, if new features are identified after the writing of this protocol, patients can be enrolled with the approval of two members of the study committee.
* Additional Criteria for Bulky Disease (lymphomas)

  * If stable disease is best response, the largest residual nodal mass must < 5 cm (approximately)
  * If response to previous therapy, the largest residual mass must represent a 50% reduction and be < 7.5 cm (approximately)
* Organ Function Criteria

Adequate organ function is defined as:

* Cardiac: Absence of decompensated congestive heart failure, or uncontrolled arrhythmia and left ventricular ejection fraction > 40%. For children that are not able to cooperate with MUGA and echocardiography, such should be clearly stated in the physician's note.
* Pulmonary: DLCO, FEV1, FVC ≥ 40% predicted, and absence of O2 requirements. For children that are not able to cooperate with PFTs, a pulse oximetry with exercise should be attempted. If neither test can be obtained it should be clearly stated in the physician's note.
* Liver: Transaminases ≤ 5 x upper limit of normal (ULN) and total bilirubin ≤ 2.5 mg/dL except for patients with Gilbert's syndrome or hemolysis
* Renal: Creatinine ≤ 2.0 mg/dl (adults) and creatinine clearance ≥ 40 mL/min (pediatrics). Adults with a creatinine > 1.2 mg/dl or a history of renal dysfunction must have estimated creatinine clearance ≥ 40 ml/min/1.73m^2. Adequate performance status is defined as Karnofsky score ≥ 70% (≥ 16 years of age) or Lansky score ≥ 50 (pediatrics)

  * Sexually active females of childbearing potential and males with partners of child-bearing potential must agree to use adequate birth control during study treatment.
  * Voluntary written consent (adult or parent/guardian with presentation of the minor information sheet, if appropriate)

Exclusion Criteria:

* Pregnant or breast feeding. The agents used in this study include Pregnancy Category D: known to cause harm to a fetus. Females of childbearing potential must have a negative pregnancy test prior to starting therapy.
* Untreated active infection
* Active HIV infection or known HIV positive serology
* Less than 3 months since prior myeloablative transplant
* Evidence of progressive disease by imaging modalities or biopsy - persistent PET activity, though possibly related to lymphoma, is not an exclusion criterion in the absence of CT changes indicating progression.
* CML in blast crisis
* Large cell lymphoma, mantle cell lymphoma and Hodgkin disease that is progressing on salvage therapy.
* Active central nervous system malignancy

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2023-02-22 (Actual); Study Completion 2024-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret MacMillan, MD, MSC, Principal Investigator — University of Minnesota
Locations (1):
- Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | No Anti-thymocyte Globulin (ATG) | Anti-thymocyte Globulin (ATG)
Started | 5 | 10
Completed | 5 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Anti-thymocyte Globulin (ATG) | Anti-thymocyte Globulin (ATG) | Total
Number analyzed (Participants) | 5 | 10 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 5 | 9 | 14
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 4 | 6 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 3 | 8 | 11
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 0 | 0 | 0
  White | 3 | 8 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 5 | 10 | 15

OUTCOME MEASURES:

1. Primary Outcome: Probability of Acute Graft Versus Host Disease (GVHD)
Description: Simple proportions will be used to estimate the probability of grade II-IV actue GVHD.
Time Frame: Day 100
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | No Anti-thymocyte Globulin (ATG) | Anti-thymocyte Globulin (ATG)
Number analyzed (Participants) | 5 | 10
Percent of participants | 0 [0 to 100] | 30 [3 to 57]

2. Secondary Outcome: Incidence of Acute GVHD
Description: Percentage of patients with grade III-IV acute GVHD.
Time Frame: Day 100
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | No Anti-thymocyte Globulin (ATG) | Anti-thymocyte Globulin (ATG)
Number analyzed (Participants) | 5 | 10
Percent of participants | 0 [0 to 100] | 10 [0 to 28]

3. Secondary Outcome: Transplant Related Mortality
Time Frame: 6 months post transplant
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | No Anti-thymocyte Globulin (ATG) | Anti-thymocyte Globulin (ATG)
Number analyzed (Participants) | 5 | 10
Percent of participants | 20 [0 to 50] | 20 [0 to 44]

4. Secondary Outcome: Chimerism
Description: Percentage of subjects with donor chimerism.
Time Frame: Day 21
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | No Anti-thymocyte Globulin (ATG) | Anti-thymocyte Globulin (ATG)
Number analyzed (Participants) | 5 | 10
Percentage of participants | 64 [0 to 81] | 89 [0 to 100]

5. Secondary Outcome: Chimerism
Description: Percentage of subjects with donor chimerism.
Time Frame: Day 100
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | No Anti-thymocyte Globulin (ATG) | Anti-thymocyte Globulin (ATG)
Number analyzed (Participants) | 5 | 8
Percentage of participants | 100 [0 to 100] | 100 [70 to 100]

6. Secondary Outcome: Chimerism
Description: Percentage of subjects with donor chimerism.
Time Frame: Day 180
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | No Anti-thymocyte Globulin (ATG) | Anti-thymocyte Globulin (ATG)
Number analyzed (Participants) | 4 | 8
Percentage of participants | 43 [0 to 100] | 100 [0 to 100]

7. Secondary Outcome: Chimerism
Description: Percentage of subjects with donor chimerism.
Time Frame: 1 year post transplant
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | No Anti-thymocyte Globulin (ATG) | Anti-thymocyte Globulin (ATG)
Number analyzed (Participants) | 3 | 8
Percentage of participants | 20 [0 to 100] | 100 [0 to 100]

8. Secondary Outcome: Neutrophil Engraftment
Description: Percentage of subjects with neutrophil engraftment.
Time Frame: Day 42
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | No Anti-thymocyte Globulin (ATG) | Anti-thymocyte Globulin (ATG)
Number analyzed (Participants) | 5 | 10
Percentage of participants | 80 [42 to 99] | 90 [64 to 99]

ADVERSE EVENTS:
Time Frame: 6 months
Description: Adverse event and/or serious adverse event recorded according to targeted reporting outlined in protocol.
  1. Events requiring prompt reporting including, but not limited to unanticipated death of a locally enrolled subject(s); new or increased risk; any adverse event that require a change to the protocol or consent form or any protocol deviation that resulting in harm
  2. graft failure by Day 42 post-transplant
Arm/Group | No Anti-thymocyte Globulin (ATG) | Anti-thymocyte Globulin (ATG)
All-Cause Mortality (participants affected / at risk) | 1/5 | 2/10
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/10
Other Adverse Events (participants affected / at risk) | 0/5 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-25): https://cdn.clinicaltrials.gov/large-docs/68/NCT02722668/Prot_SAP_000.pdf
  • Informed Consent Form (2022-04-25): https://cdn.clinicaltrials.gov/large-docs/68/NCT02722668/ICF_001.pdf